CLINICAL TRIAL: NCT01313949
Title: Peer Leaders Accelerated Training Initiative to Unleash Potential of Mentorship (PLATINUM) Program: A Feasibility Study on a Train-the-trainer Course on Peer Support for People With Type 2 Diabetes
Brief Title: PLATINUM Program: A Feasibility Study on a Train-the-trainer Course on Peer Support for People With Type 2 Diabetes
Acronym: PLATINUM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asia Diabetes Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CRE-2009-087
Record Dates: First submitted 2011-03-07; First posted 2011-03-14 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-07

CONDITIONS: Diabetes
Keywords: Diabetes; Peer Support; Structured Care
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (No Intervention): A total of 90 patients with diabetes will be recruited. Thirty will be selected for the training course and the other 60 will be compared as controls. These controls will receive their usual diabetes care.
- Peer leader training (Experimental): Peer leaders are people with diabetes who had volunteered to undertake an extensive program of training. The purpose of this training is to make them effective in the provision of support and advice to their peers on a one-to-one basis via telecommunication.
  These diabetes patients will undergo a 32-hour 'Train the trainer' program (4 workshops, 8-hours each) led by health care experts in nutrition, physical activity, psychology and neuro-linguistic program [NLP] trainer to ensure the adequacy of knowledge and skills of these mentors.
  Interventions: Other: Training program

INTERVENTIONS:
Other: Training program — These diabetes patients will undergo a 32-hour 'Train the trainer' program (4 workshops, 8-hours each) led by health care experts in nutrition, physical activity, psychology and neuro-linguistic program [NLP] trainer to ensure the adequacy of knowledge and skills of these mentors.
  Arms: Peer leader training

SUMMARY:
The investigators hypothesize that a training course to people with diabetes on peer support and empowerment will improve their glycemic parameters, knowledge on diabetes and level of self efficacy. This group of trained patients (peer leaders) should be competent to teach and help other patients with diabetes through peer support and empowerment on better self management of their diabetes.

DETAILED DESCRIPTION:
In our attempt to improve diabetes self care, one important component is the diabetes patients who should have the best incentive to improve their care levels and reduce their complication risk, provided that they are appropriately trained, informed, educated and supported. According to the World Health Organization (WHO) Innovative Care for Chronic Conditions framework, expert patients are recommended to be included in the health care team to make them prepared, motivated and informed decision makers to preserve health and improve clinical outcomes. In a recent report on WHO consultation, peer support interventions are considered to have enormous potentials to make self management an effective component of chronic care.

Peer support is defined as support from a person who has experiential knowledge of a specific behavior or stressor and similar characteristics as the target population. Thus people with common illness experience can share knowledge and experience in a less hierarchical and reciprocal relationship compared to that between patients and health care professionals. A number of programs including health worker-led groups with peer exchange, peer-led face-to-face self management programs, peer coaches and remote peer support have reported encouraging results with short term improvement in metabolic or cognitive-psychological-behavioral dimensions, although these results are often limited by non-sustainability of changes and insufficient reach or adoption of programs by patients or health care workers. In the WHO report, health care experts from various disciplines concluded that whilst peer support is a promising approach for diabetes management, issues regarding methods of organization, types of programs and their integration with other clinical and outreach services remain to be addressed. Of note, there is a paucity of similar data in developing and low income areas which are hit hardest by this epidemic and where peer support program may offer great promise to make diabetes prevention and care program more sustainable and accessible, if implemented and evaluated systematically.

Health professionals, especially diabetes nursing specialists, have been training diabetes patients on the understanding and self-caring of diabetes. However, with the emerging concept and preliminary evidence of success in the role of "peer advisors" in diabetes to lead self care courses for other fellow patients, a train-the-trainer program to develop "expert patients" is essential. On top of factual knowledge on diabetes as a disease, context of this program needs to cover include communication and empowerment skill, basic knowledge on psychology, stress management, social support, empowerment, healthy lifestyle including diet and physical activity.

In the evaluation of the programs, there is a need to define the qualities and roles of the peer supporter, design programs which integrate and complement formal health services, identify optimal mix of modalities of intervention, types and dose response of these interventions and evaluate acceptability and effectiveness of these programs in different cultures. Other evaluation indexes include effects of programs on behavioral changes, knowledge and attitudes, functionality, clinical care as well as their cost effectiveness, reach, implementation-consistency, adoption and maintenance of effects over time.

ELIGIBILITY:
Inclusion Criteria:

* Chinese people with type 2 diabetes
* 18-75 years of age
* Good glycaemic control (HbA1c <7%) and remain stable in past 1 year
* Willing to complete the structured training curriculum to prepare themselves as peer leaders
* Fluent in Cantonese

Exclusion Criteria:

* Known psychiatric disease
* Physically handicapped to the degree that communication with others is significantly impaired impaired, such as deafness, paraplegia.
* Illiterate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2009-02; Primary Completion 2011-02 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
To assess the effectiveness of the training program in improving glycemic parameters in diabetic patients before and after the training. | 6 months
  Metabolic parameters, such as HbA1c, Body Mass Index (BMI), Lipid Profile, etc. will be measured at specific time points before and after the training

SECONDARY OUTCOMES:
To assess the efficacy of the training on the attitudes, behaviours and self-efficacy of the participants as compared to the control patients | 6 months
  The psychosocial-behavior assessment will include using the Summary of Diabetes Self- Care Activities (SDSCA), Diabetes Empowerment Scale (DES), Depression Anxiety Stress Scale-21 (DASS21), General Health Questionnaire (GHQ12), Euro Quality of Life (EQ5D) & Patient Health Questionniare (PHQ9).
To assess the efficacy of the training in improving the participants' knowledge of diabetes, as compared to the control patients. | 6 months
  An evaluation feedback form will be completed by all participants after each workshop

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Wong, Principal Investigator — Prince of Wales Hospital, Shatin, HK; Shimen Au, Principal Investigator — Ruttonjee & Tang Shiu Kin Hospitals, Wan Chai, HK
Locations (15):
- Hong Kong (15):
  - Diabetes Ambulatory Care Centre, UCH, Kwun Tong, Kowloon
  - Kwai Chung out-patient clinic, Kwai Chung, New Territories
  - CUHK YCK, Prince of Wales Hospital, Shatin, New Territories
  - Diabetes & Endocrine Centre, Prince of Wales Hospital, Shatin, New Territories
  - Diabetes Centre, North District Hospital, Sheung Shui, New Territories
  - Diabetes Centre, Tung Wah Eastern Hospital, Causeway Bay
  - Diabetes Hong Kong, Central
  - Diabetes Ambulatory Centre, PYNEH, Chai Wan
  - Diabetes Centre, Kwong Wah Hospital, Kowloon
  - Diabetes Centre, Queen Elizabeth Hospital, Kowloon
  - PMH, Diabetes Care Centre, Princess Margaret Hospital, Kowloon
  - Lam Tin Health Clinic, Lam Tin
  - Diabetes Centre, Queen Mary Hospital, Pok Fu Lam
  - Sai Wan Ho Health Centre, Sai Wan Ho
  - Diabetes Centre, Ruttonjee Hospital, Wan Chai

REFERENCES:
- See also: For more information on this trial and others conducted by the Asia Diabetes Foundation. — http://www.adf.org.hk